CLINICAL TRIAL: NCT00403624
Title: Clinical Study to Evaluate a Protocol of Oxaliplatin -UFT- Radiotherapy for the Neoadjuvant Treatment Rectal Cancer
Brief Title: Evaluation of the Neoadjuvant Treatment With Oxaliplatin -UFT- Radiotherapy in Rectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8128
Record Dates: First submitted 2006-11-23; First posted 2006-11-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-04

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: OXALIPLATIN

SUMMARY:
Primary objective:

- To evaluate the rate of responses to neoadjuvant therapy + radiotherapy

Secondary objective:

- tolerability (toxicity) and time to progression

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* Patients with measurable, histologically proven rectal cancer.
* No history of previous malignancy but adequately treated skin / cervical cancer.
* Adequate haematological, renal and liver function.

Exclusion Criteria:

* No cardiopulmonary insufficiency or coronary disease. No sensory neuropathy prior to study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2001-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Tumour response

SECONDARY OUTCOMES:
Disease free and Overall survival ; Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Dr., Study Director — Sanofi